CLINICAL TRIAL: NCT02245542
Title: The Impact of Alna® Ocas® on Nocturia in Patients With Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia (LUTS/BPH)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.68
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- BPH patients
  Interventions: Drug: ALNA®OCAS®

INTERVENTIONS:
Drug: ALNA®OCAS®

SUMMARY:
Study to assess efficacy, tolerability and safety parameters of a three month ALNA®OCAS® -treatment with special respect to nocturia

ELIGIBILITY:
Inclusion Criteria:

* Indication for treatment with ALNA®OCAS® according to the prescribing information for a minimum period of three months

Exclusion Criteria:

* Patients fulfilling one of the general or specific contraindications listed in the ALNA®OCAS® Summary of Product Characteristics (SPC), particularly patients with known hypersensitivities against tamsulosin hydrochloride or any other ingredient of the product, orthostatic dysregulation or severe liver insufficiency could not be included in the Post Marketing Study (PMS) study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BPH patients who are indicated for treatment with ALNA®OCAS® with special respect to nocturia recruited at urologists
Sampling Method: Non-Probability Sample
Enrollment: 5775 (Actual)
Dates: Start 2005-04; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in International Prostatic Symptom Score (IPSS) by means of a patient questionnaire | Baseline, after 3 months
Change from Baseline in Nocturia quality of life by means of a patient questionnaire | Baseline, after 3 months

SECONDARY OUTCOMES:
Change from Baseline in Maximum urinary flow rate (Qmax) | Baseline, after 3 months
Change from Baseline in residual urine volume | Baseline, after 3 months
Assessment of tolerability by investigator on 4-point scale | after 3 months
Number of patients with adverse events | up to 3 months